CLINICAL TRIAL: NCT06555783
Title: A Phase 2, Parallel-Group, Dose-Range-Finding Study With Randomized Double-Blind Treatment and Open-Label Periods to Evaluate the Safety and Efficacy of ALKS 2680 in Subjects With Narcolepsy Type 2
Brief Title: A Study to Evaluate the Safety and Effectiveness of ALKS 2680 in Subjects With Narcolepsy Type 2
Acronym: Vibrance-2
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alkermes, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ALKS 2680-202
Record Dates: First submitted 2024-08-13; First posted 2024-08-15 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Narcolepsy Type 2
Keywords: Narcolepsy; Narcolepsy Type 2; NT2; Orexin-2 receptor agonist; Sleep; Sleep disorder; Excessive daytime sleepiness
MeSH Terms: conditions — Narcolepsy; Sleep Wake Disorders; Disorders of Excessive Somnolence

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (4):
- ALKS 2680, 10 mg (Experimental): Oral tablet containing 10mg of ALKS 2680 for once daily administration
  Interventions: Drug: ALKS 2680
- ALKS 2680, 14 mg (Experimental): Oral tablet containing 14mg of ALKS 2680 for once daily administration
  Interventions: Drug: ALKS 2680
- ALKS 2680, 18 mg (Experimental): Oral tablet containing 18mg of ALKS 2680 for once daily administration
  Interventions: Drug: ALKS 2680
- Placebo (Placebo Comparator): Oral tablet containing matching placebo for once daily administration
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ALKS 2680 — Oral tablet containing ALKS 2680
  Arms: ALKS 2680, 10 mg; ALKS 2680, 14 mg; ALKS 2680, 18 mg
Drug: Placebo — Oral tablet containing placebo for once daily administration
  Arms: Placebo

SUMMARY:
The purpose of this study is to measure the safety and decrease in sleepiness in subjects with narcolepsy type 2 (NT2) when taking ALKS 2680 tablets compared to placebo tablets.

ELIGIBILITY:
Inclusion Criteria:

* 18-70 years of age
* Has a BMI ≥18 and ≤40 kg/m2
* Meets the diagnostic criteria of Narcolepsy type 2 according to ICSD-3-TR guidelines.

Additionally, meets the following criteria:

* Has residual excessive daytime sleepiness
* Is willing and able to discontinue any medications prescribed for the management of narcolepsy symptoms for at least 14 days and for the duration of study
* Is willing to adhere to additional protocol requirements

Exclusion Criteria:

* Significant comorbid medical conditions, including other sleep, cardiovascular, psychiatric, hepatic or other disorders may be exclusionary; eligibility will be determined on an individual basis by the study investigator
* Is currently pregnant, breastfeeding, or planning to become pregnant during the study
* Is currently enrolled in another clinical study (other than the parent study) or used any investigational drug or device within 30 days prior to Screening

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2024-07-26 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in Mean Sleep Latency (MSL) on the Maintenance Wakefulness Test (MWT) | Baseline to Week 8
Change in Epworth Sleepiness Scale (ESS) | Baseline to week 8
  Participants will be asked to complete the ESS, reporting on the level of sleepiness they experienced over the past 7 days.

SECONDARY OUTCOMES:
Incidence of adverse events | Up to 21 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, MD, Study Director — Alkermes, Inc.
Locations (45):
- United States (32):
  - Alkermes Investigator Site, Little Rock, Arkansas
  - Alkermes Investigator Site, Los Angeles, California
  - Alkermes Investigator Site, Redwood City, California
  - Alkermes Investigator Site, San Francisco, California
  - Alkermes Investigator Site, Santa Ana, California
  - Alkermes Investigational Site, Aurora, Colorado
  - Alkermes Investigator Site, Colorado Springs, Colorado
  - Alkermes Investigator Site, Brandon, Florida
  - Alkermes Investigator Site, Miami, Florida
  - Alkermes Investigator Site, Winter Park, Florida
  - Alkermes Investigator Site, Atlanta, Georgia
  - Alkermes Investigational Site, Macon, Georgia
  - Alkermes Investigator Site, Stockbridge, Georgia
  - Alkermes Investigational Site, Peoria, Illinois
  - Alkermes Investigator Site, Lansing, Michigan
  - Alkermes Investigator Site, Sterling Heights, Michigan
  - Alkermes Investigator Site, Lincoln, Nebraska
  - Alkermes Investigator Site, Middletown, New Jersey
  - Alkermes Investigator Site, Denver, North Carolina
  - Alkermes Investigator Site, Huntersville, North Carolina
  - Alkermes Investigator Site, Canton, Ohio
  - Alkermes Investigator Site, Cincinnati, Ohio
  - Alkermes Investigational Site, Cleveland, Ohio
  - Alkermes Investigator Site, Abington, Pennsylvania
  - Alkermes Investigational Site, Philadelphia, Pennsylvania
  - Alkermes Investigator Site, Wyomissing, Pennsylvania
  - Alkermes Investigator Site, Columbia, South Carolina
  - Alkermes Investigator Site, Austin, Texas
  - Alkermes Investigator Site, San Antonio, Texas
  - Alkermes Investigational Site, Sugar Land, Texas
  - Alkermes Investigator Site, Sugarland, Texas
  - Alkermes Investigational Site, Madison, Wisconsin
- Australia (2):
  - Alkermes Investigator Site, Macquarie Park, New South Wales
  - Alkermes Investigator Site, Bedford Park, South Australia
- Belgium (2):
  - Alkermes Investigational Site, Alken
  - Alkermes Investigational Site, Namur
- Alkermes Investigational Site, Prague, Czechia
- France (2):
  - Alkermes Investigational Site, Bordeaux, Bordeaux
  - Alkermes Investigational Site, La Tronche, LA Tronche
- Italy (3):
  - Alkermes Investigational Site, Bologna, BO
  - Alkermes Investigational Site, Milan, Metropolitan City of Milan
  - Alkermes Investigational site, Verona
- Alkermes Investigational Site, Zwolle, Netherlands
- Spain (2):
  - Alkermes Investigational Site, Barcelona
  - Alkermes Investigational Site, Madrid

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Vibrance-2 Study — https://vibrancestudies.com/?utm_source=ClinicalTrials&utm_medium=Referral&utm_content=Listing&utm_campaign=Listing_Vibrance2